CLINICAL TRIAL: NCT05033041
Title: Comparison of Gastric Volumes by Gastric Ultrasound in Term Parturients Undergoing Scheduled Elective Cesarean Delivery With and Without Metoclopramide
Brief Title: Gastric Volumes by US in Term Parturients Undergoing CS With and Without Metoclopramide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jennifer Banayan, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00215570
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy; Cesarean Section; Aspiration
Keywords: Pregnancy; Gastric Volume; Ultrasound Measurement; Aspiration Prevention; Cesarean Section

STUDY DESIGN:
Intervention Model Description: Randomized controlled blinded study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research pharmacy to prepare the study medication blinding the participant, care providers, investigator and outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 Study Drug Metoclopramide (Active Comparator): Intravenous administration of 10 mg metoclopramide
  Interventions: Drug: Study drug metoclopramide
- Group 2 Study Drug Placebo (Placebo Comparator): Intravenous administration of sterile normal saline
  Interventions: Drug: Study drug placebo administration

INTERVENTIONS:
Drug: Study drug metoclopramide — Intravenous administration of 10 mg metoclopramide
  Arms: Group 1 Study Drug Metoclopramide
Drug: Study drug placebo administration — Intravenous administration of placebo (sterile normal saline)
  Arms: Group 2 Study Drug Placebo

SUMMARY:
Our objective is to compare gastric volumes (mL) between women who receive metoclopramide versus placebo prior to scheduled cesarean delivery in appropriately fasted patients. If metoclopramide is found not to reduce gastric volumes this would inform future practice guidelines for obstetric anesthesia, which currently recommends metoclopramide administration prior to cesarean deliveries.

We hypothesize that metoclopramide given to women with appropriate fasting prior to cesarean delivery does not result in any clinically significant reduction in gastric volume (mL) and therefore does not provide any additional benefit for aspiration prophylaxis but may expose patients to unnecessary side effects. A secondary objective will be to evaluate if gastric volume is a significant predictor of intraoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (ASA Physical Status 2)
* Age >18 years old
* Non-obese (BMI <40 kg/m2)
* Age >18 years
* Term (>37 week)
* Non-laboring parturient
* Single gestation
* Scheduled for a cesarean delivery and NPO

Exclusion Criteria:

* Systemic disease such as diabetes mellitus (type 1 or 2)
* Multiple gestation
* Abnormality of upper GI tract
* History of GI tract related surgical procedures
* Use of gastric motility medications
* Active labor
* Renal impairment (creatinine >2)
* Non-English speaking
* Cognitively impaired
* History of QT prolongation
* Use of general anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant undergoing cesarean section.
Enrollment: 72 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Banayan, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital and Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] MENDELSON CL. The aspiration of stomach contents into the lungs during obstetric anesthesia. Am J Obstet Gynecol. 1946 Aug;52:191-205. doi: 10.1016/s0002-9378(16)39829-5. No abstract available. PMID 20993766
- [Background] Practice Guidelines for Obstetric Anesthesia: An Updated Report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia and the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2016 Feb;124(2):270-300. doi: 10.1097/ALN.0000000000000935. No abstract available. PMID 26580836
- [Background] 4. Knight M, Bunch K, Tuffnell D, Shakespeare J, Kotnis R, Kenyon S, Kurinczuk JJ (Eds.) on behalf of MBRRACE-UK. Saving Lives, Improving Mothers' Care - Lessons learned to inform maternity care from the UK and Ireland Confidential Enquiries into Maternal Deaths and Morbidity 2016-18. Oxford: National Perinatal Epidemiology Unit, University of Oxford 2020.
- [Background] Leus M, van de Ven A. IMAGES IN CLINICAL MEDICINE. An Acute Dystonic Reaction after Treatment with Metoclopramide. N Engl J Med. 2015 Oct;373(14):e16. doi: 10.1056/NEJMicm1412207. No abstract available. PMID 26422744
- [Background] Mishriky BM, Habib AS. Metoclopramide for nausea and vomiting prophylaxis during and after Caesarean delivery: a systematic review and meta-analysis. Br J Anaesth. 2012 Mar;108(3):374-83. doi: 10.1093/bja/aer509. Epub 2012 Feb 3. PMID 22307240
- [Background] Paranjothy S, Griffiths JD, Broughton HK, Gyte GM, Brown HC, Thomas J. Interventions at caesarean section for reducing the risk of aspiration pneumonitis. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD004943. doi: 10.1002/14651858.CD004943.pub3. PMID 20091567
- [Background] Perlas A, Mitsakakis N, Liu L, Cino M, Haldipur N, Davis L, Cubillos J, Chan V. Validation of a mathematical model for ultrasound assessment of gastric volume by gastroscopic examination. Anesth Analg. 2013 Feb;116(2):357-63. doi: 10.1213/ANE.0b013e318274fc19. Epub 2013 Jan 9. PMID 23302981
- [Background] Van de Putte P, Perlas A. Ultrasound assessment of gastric content and volume. Br J Anaesth. 2014 Jul;113(1):12-22. doi: 10.1093/bja/aeu151. Epub 2014 Jun 3. PMID 24893784
- [Background] Arzola C, Perlas A, Siddiqui NT, Carvalho JCA. Bedside Gastric Ultrasonography in Term Pregnant Women Before Elective Cesarean Delivery: A Prospective Cohort Study. Anesth Analg. 2015 Sep;121(3):752-758. doi: 10.1213/ANE.0000000000000818. PMID 26097988
- [Background] Arzola C, Perlas A, Siddiqui NT, Downey K, Ye XY, Carvalho JCA. Gastric ultrasound in the third trimester of pregnancy: a randomised controlled trial to develop a predictive model of volume assessment. Anaesthesia. 2018 Mar;73(3):295-303. doi: 10.1111/anae.14131. Epub 2017 Dec 19. PMID 29265187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 72 Subjects were randomized to treatment.
Groups:
- Group 1 Study Drug Metoclopramide: Intravenous administration of 10 mg metoclopramide
  Study drug metoclopramide: Intravenous administration of 4 mg metoclopramide
Period: Overall Study
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Started | 38 | 34
Completed | 38 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo | Total
Number analyzed (Participants) | 38 | 34 | 72
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 35 [33 to 38] | 35 [32 to 39] | 35 [32 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 34 | 72
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 31 | 31 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 36 | 32 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 34 | 72
Weight (kg) [Median (Inter-Quartile Range); unit: Kilograms] | 80.5 [73.3 to 86] | 79.5 [73.3 to 86] | 80 [73.3 to 86]
Body Mass In kg/m^2 [Median (Inter-Quartile Range); unit: kg/m^2] | 29.8 [27.4 to 31.8] | 29.6 [26.2 to 33.1] | 29.7 [26.2 to 33.1]
Gestational age (weeks) [Median (Inter-Quartile Range); unit: Weeks] | 39.1 [39 to 39.2] | 39.1 [39 to 39.3] | 39.1 [39 to 39.3]
Gravid (number of pregnancies) [Count of Participants; unit: Participants]
  Gravid 1 | 9 | 3 | 12
  Gravid 2 | 12 | 16 | 28
  Gravid 3 | 6 | 8 | 14
  Greater or equal to gravid 4 | 11 | 7 | 18
Parity [Count of Participants; unit: Participants]
  0 | 12 | 4 | 16
  1 | 21 | 22 | 43
  2 | 5 | 5 | 10
  Greater or equal to 3 | 0 | 3 | 3
Prior cesarean deliveries [Count of Participants; unit: Participants] — Number of participants who have had a previous cesarean delivery.
  Participants | 25 | 29 | 54
Gastroesophageal reflux disease (GERD) [Count of Participants; unit: Participants]
  With pregnancy | 31 | 24 | 55
  Currently | 4 | 7 | 11
Hours since last solid ingestion (NPO) [Median (Inter-Quartile Range); unit: Hours] | 12.5 [7.5 to 13.7] | 12.9 [8.3 to 14.6] | 12.7 [7.5 to 14.6]
Time from last liquid ingestion (hours) [Median (Inter-Quartile Range); unit: Hours] | 3.3 [3 to 3.7] | 3.4 [3 to 4.4] | 3.3 [3 to 4.4]
Pretreatment estimated gastric volume (mL) [Median (Inter-Quartile Range); unit: Milliliters]
  Perlas calculation | 41 [32 to 53] | 43 [32 to 52] | 42 [32 to 53]
  Roukhomovsky calculation | 53 [40 to 81] | 53 [40 to 75] | 53 [40 to 81]

OUTCOME MEASURES:

1. Primary Outcome: Change in Gastric Volume (mL)
Description: Change in gastric volume (mL) determined by gastric ultrasound before and 30 minutes after administration of study drug. Gastric volumes were calculated from the cross sectional area (CSA) area using both the Perlas (Volume=27.0+14.6*(RLD CSA (cm2)-1.28 * age)) and the Roukhomovsky method (volume=(0.18*RLD CSA (mm2))+(0.11*SUP CSA (mm2)-62.4) methods.
Time Frame: 30 minutes after administration of study drug
Population: One subject in the placebo group did not have a paired ultrasound (missing pre-treatment).
Measure: Median (95% Confidence Interval); unit: Milliliters
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 33
Milliliters
  Perlas method | -1 [-8 to 6] | -2 [-7 to 3]
  Roukhomovsky formula | 0 [-10 to 9] | 1 [-6 to 6]
Statistical Analysis 1: Comparison: Group 1 Study Drug Metoclopramide vs Group 2 Study Drug Placebo; Comparison of the means using two one-sided t tests (TOST); Test type: Equivalence — Equivalence is based on an equivalence hypothesis of -17mL <difference in differences < 17mL; p = .001, t-test, 1 sided

2. Secondary Outcome: Subject Report of Nausea During Cesarean Section
Description: Subject reported intraoperative nausea during the cesarean delivery
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Participants | 14 | 18

3. Secondary Outcome: Adverse Events
Description: Number of reported adverse events experienced for each group.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Participants
  Akathisia | 0 | 0
  Extrapyramidal effect | 0 | 0
  High fever | 0 | 0
  Muscle stiffness | 0 | 0
  Depression | 0 | 0
  Fluid retention | 0 | 0
  Hypoprolactinemia | 0 | 0
  Hypersensitivity reaction | 0 | 0
  Blood cell changes | 0 | 0
  Hypernatremia | 0 | 0
  Maternal resuscitation | 0 | 0
  Maternal hypertension | 1 | 1
  Infant gastrointestinal disturbances | 0 | 0
  Infant extrapyramidial effects | 0 | 0
  Infant methemoglobinemia | 0 | 0

4. Secondary Outcome: Intraoperative Nausea Occurrences
Description: Number of nausea occurrences during cesarean section procedure
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: Nausea occurrences
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Nausea occurrences | 1 [1 to 1] | 2 [1 to 4]

5. Secondary Outcome: Intraoperative Nausea Time From Intrathecal Anesthesia to Nausea Episode in Minutes
Description: Total elapsed time in minutes from the placement of the intrathecal medications by anesthesiology team to the first experience of nausea reported by the participant.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Minutes | 26 [4 to 51] | 20 [7 to 28]

6. Secondary Outcome: Subject Experienced Vomiting During Cesarean Section
Description: Subject experienced vomiting episode during the cesarean delivery procedure.
Time Frame: 24 Hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Participants | 3 | 5

7. Secondary Outcome: Number of Intraoperative Vomiting Occurrences
Description: Number of intraoperative vomiting occurrences during the cesarean section.
Time Frame: 24 Hours
Measure: Median (Inter-Quartile Range); unit: Number of episodes
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Number of episodes | 1 [1 to 2] | 1 [1 to 2]

8. Secondary Outcome: Time From Intrathecal Anesthesia to Vomiting Episode in Minutes.
Description: The elapsed time in minutes from anesthesia team placing the intrathecal medications to the first episode of vomiting during.
Time Frame: 24 Hours
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Minutes | 34 [8 to 34] | 26 [22 to 34]

9. Secondary Outcome: Antiemetic Prophylaxis
Description: Subject received antiemetic prophylaxis of ondansetron or dexamethasone prior to the cesarean section.
Time Frame: 24 Hours
Measure: Number; unit: participants
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
participants
  Received ondansetron | 35 | 32
  Received dexamethasone | 34 | 32

10. Secondary Outcome: PACU Antiemetic Treatment (n)
Description: Number of participants who required antiemetic medications in the post anesthesia care unit
Time Frame: 24 hours
Measure: Number; unit: Participants
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Participants | 5 | 1

11. Secondary Outcome: Nausea After PACU Discharge
Description: Number of participants who experienced nausea after being discharged from the post anesthesia care unit
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Participants | 3 | 6

12. Secondary Outcome: Elapsed Time From Study Drug to Second Ultrasound
Description: Total elapsed time in minutes after study drug administered to second gastric ultrasound.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Minutes | 30 (1) | 30 (2)

13. Secondary Outcome: Second Ultrasound Cross Sectional Area (cm^2)
Description: The cross sectional area in centimeters squared for the second gastric ultrasound which was performed 30 minutes after study medication administered
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: Centimeters
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Centimeters
  Supine position | 3.7 [3.1 to 4.4] | 3.5 [3.1 to 4.3]
  Right lateral displacement position | 4.0 [3.6 to 5.0] | 4 [3.4 to 5.2]

14. Secondary Outcome: Post Treatment Estimated Volume (mL) Second Ultrasound
Description: Gastric volume in milliliters of the second ultrasound obtained 30 minutes after study drug administration
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: Milliliters
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Milliliters
  Perlas calculation | 43 [32 to 55] | 39 [32 to 59]
  Roukhomovsky calculation | 55 [38 to 75] | 54 [36 to 72]

15. Secondary Outcome: Second Ultrasound Volume >1.5 * Weight (kg)
Description: Number of subjects experiencing a volume greater than than 1.5 times weight in kilograms after the second gastric ultrasound 30 minutes after study medication administration.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Participants
  Perlas calculation | 0 | 0
  Roukhomovsky calculation | 2 | 3

16. Other Pre Specified Outcome: First Ultrasound Stomach Cross-sectional Area (cm2)
Description: The first ultrasound of the stomach cross-sectional area in centimeters squared.
Time Frame: After consent obtained
Measure: Median (Inter-Quartile Range); unit: centimeters squared
Units Other Than Participants: Ultrasounds
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Number analyzed (Ultrasounds) | 38 | 34
centimeters squared
  Supine | 3.8 [3.0 to 4.5] | 3.6 [3.3 to 4.4]
  Right lateral displacement | 3.9 [3.3 to 4.9] | 4.1 [3.3 to 5.0]

17. Other Pre Specified Outcome: First Ultrasound Volume Greater Than 1.5 * Weight (kg)
Description: The first ultrasound calculated volume greater than 1.5 times weight in kilograms.
Time Frame: After consent obtained
Measure: Number; unit: participants
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
participants
  Perlas calculation | 0 | 0
  Roukhomovsky calculation | 2 | 2

18. Post Hoc Outcome: Neonatal Outcome APGAR Score
Description: Neonatal APGAR scores at 1 and 5 minutes (0-poor 10 good)
Time Frame: 5 minutes after delivery
Measure: Median (Inter-Quartile Range); unit: scores on a scale (0 poor-10 good)
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
scores on a scale (0 poor-10 good)
  1 Minute APGAR score | 8 [8 to 9] | 8.5 [8 to 9]
  5 Minute APGAR score | 9 [9 to 9] | 9 [9 to 9]

19. Post Hoc Outcome: Neonatal Outcomes Arterial Blood Gasses
Description: Neonatal arterial blood gas results obtained at delivery (pH).
Time Frame: 5 minutes after delivery
Measure: Median (Inter-Quartile Range); unit: pH
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
pH | 7.25 [7.22 to 7.29] | 7.25 [7.22 to 7.29]

20. Post Hoc Outcome: Neonatal Outcomes Venous Blood Gas
Description: Neonatal venous blood gas post delivery (pH)
Time Frame: 5 minutes after delivery
Measure: Median (Inter-Quartile Range); unit: pH
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
pH | 7.30 [7.28 to 7.34] | 7.32 [7.29 to 7.34]

21. Post Hoc Outcome: Neonatal Outcomes: Neonatal Resuscitation
Description: Neonate required neonatal resuscitation required after cesarean section delivery
Time Frame: 24 hours
Measure: Number; unit: Participants
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Participants | 11 | 9

22. Post Hoc Outcome: Neonatal Outcomes: NICU Admission
Description: Neonate admission to the newborn intensive care unit
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
Participants | 2 | 0

23. Post Hoc Outcome: Neonatal Outcomes Arterial Blood Gasses
Description: Neonatal arterial blood gas results obtained at delivery (O2 (mmHg), CO2 (mmHg).
Time Frame: After delivery
Measure: Median (Inter-Quartile Range); unit: millimeters of mercury
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
millimeters of mercury
  Arterial blood gas 02 (mmHg) | 27 [19 to 60] | 32 [21 to 62]
  Arterial blood gas C02 (mmHg) | 57 [50 to 60] | 56 [47 to 61]

24. Post Hoc Outcome: Neonatal Outcomes Venous Blood Gas
Description: Neonatal venous blood gas post delivery including pH, O2 (mmHg), C02 (mmHg)
Time Frame: After delivery
Measure: Median (Inter-Quartile Range); unit: millimeters of mercury
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
Number analyzed (Participants) | 38 | 34
millimeters of mercury
  Venous blood gas oxygen (mmHg) | 36 [27 to 49] | 41 [29 to 53]
  Venous blood gas C02 (mmHg) | 44 [41 to 49] | 45 [42 to 48]

ADVERSE EVENTS:
Time Frame: 72 Hours
Arm/Group | Group 1 Study Drug Metoclopramide | Group 2 Study Drug Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/34
Other Adverse Events (participants affected / at risk) | 3/38 | 6/34
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Study Drug Metoclopramide (N=38) | Group 2 Study Drug Placebo (N=34)
Nausea (Gastrointestinal disorders) | 3 (3) | 6 (6)
Hypertension (Blood and lymphatic system disorders) | 3 (3) | 6 (6) — Hypertension during hospitalization for delivery of baby

LIMITATIONS AND CAVEATS:
We recognize the potential limitations that some providers may still choose to administer metoclopramide to augment esophageal contractions despite its limited impact on esophageal junction compliance. While metoclopramide may help augment contractions, its use in fasted patients who are at low risk of gastric contents >1.5mL/kg is unlikely to significantly impact aspiration risk, making its benefit in this context less clear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT05033041/Prot_SAP_000.pdf